CLINICAL TRIAL: NCT02149875
Title: A Comparison of Safety and Efficacy of Dl-3-n-butylphthalide and Cerebrolysin on Neurological and Behavioral Outcomes in Acute Ischemic Stroke: a Randomized, Double-blind Study.
Brief Title: Dl-3-n-butylphthalide and Cerebrolysin Treatment in Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, Doctor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 605872
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Acute Cerebral Stroke Within 12 Hours for the First Time
Keywords: Acute ischemic stroke; Dl-3-n-butylphthalide; Cerebrolysin
MeSH Terms: conditions — Ischemic Stroke | interventions — 3-n-butylphthalide; Long-Term Synaptic Depression; cerebrolysin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dl-3-n-butylphthalide (Experimental): Intravenous infusion of 25mg dl-3-n-butylphthalide b.i.d.for 10 days
  Interventions: Drug: Dl-3-n-butylphthalide
- Cerebrolysin (Experimental): Intravenous infusion of 30 ml cerebrolysin q.d. for 10 days
  Interventions: Drug: Cerebrolysin
- Placebo (Placebo Comparator): Intravenous infusion of 100 ml saline intravenous q.d. for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dl-3-n-butylphthalide — Intravenous infusion of 100 ml dl-3-n-butylphthalide and sodium chloride injection for 10 days, twice daily.
  Other Names: CSPC NBP Pharmaceutical Co., Ltd., Shijiazhuang, China
  Arms: Dl-3-n-butylphthalide
Drug: Cerebrolysin — Intravenous infusion of 30 ml Cerebrolysin per day in 100 ml normal saline for 10 days.
  Other Names: Ever Pharma, Unterach am Attersee, Austria
  Arms: Cerebrolysin
Drug: Placebo — 100 ml saline intravenous infusion once daily for 10 days.
  Other Names: Hebei Tiancheng Pharmaceutical Co., Ltd., Cangzhou, China
  Arms: Placebo

SUMMARY:
The investigators conducted a randomized, double-blind, trial enrolled 60 patients within 12 hours of acute ischemic stroke (AIS) in China. Patients were randomly assigned to receive a 10-day infusion of dl-3-n-butylphthalide (NBP) or cerebrolysin, or placebo. National Institutes of Health Stroke Scale (NIHSS) and Barthel Index (BI) were used to evaluate the efficacy in the patients with AIS at 11-day and 21-day after therapy. Adverse events were also analyzed among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke within 12 hours for the first time before entry into the study
* National Institutes of Health Stroke Scale (NIHSS) score between 6 and 25

Exclusion Criteria:

* with lacunar infarction
* with cerebral hemorrhagic infarction
* with epilepsy or epileptic persons
* with history of neurological diseases
* with myocardial infarction,
* with renal and hepatic abnormalities
* with metabolic diseases
* with contraindications to antiplatelet treatments

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Xue, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue LX, Zhang T, Zhao YW, Geng Z, Chen JJ, Chen H. Efficacy and safety comparison of DL-3-n-butylphthalide and Cerebrolysin: Effects on neurological and behavioral outcomes in acute ischemic stroke. Exp Ther Med. 2016 May;11(5):2015-2020. doi: 10.3892/etm.2016.3139. Epub 2016 Mar 10. PMID 27168844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2010 to May 2010, a randomized, double-blind trial was conducted, which involved patients with AIS in the Neurology Ward of Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Shanghai, China).
Groups:
- Dl-3-n-butylphthalide: Intravenous infusion of 25mg dl-3-n-butylphthalide b.i.d.for 10 days
  "Dl-3-n-butylphthalide", "Cerebrolysin" and "Placebo" separately
- Cerebrolysin: Intravenous infusion of 30 ml cerebrolysin q.d. for 10 days
  "Dl-3-n-butylphthalide", "Cerebrolysin" and "Placebo" separately
- Placebo: Intravenous infusion of 100 ml saline intravenous q.d. for 10 days
  "Dl-3-n-butylphthalide", "Cerebrolysin" and "Placebo" separately
Period: Overall Study
Arm/Group | Dl-3-n-butylphthalide | Cerebrolysin | Placebo
Started | 27 | 28 | 29
Completed | 20 | 20 | 20
Not Completed | 7 | 8 | 9
Not completed — Lost to Follow-up | 3 | 4 | 5
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Physician Decision | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dl-3-n-butylphthalide | Cerebrolysin | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (6.3) | 66.5 (8.1) | 68.4 (4.2) | 67.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 10 | 32
  Male | 9 | 9 | 10 | 28
Time until admission [Mean (Standard Deviation); unit: hour] | 5.4 (3.0) | 5.0 (3.3) | 4.8 (3.7) | 5.1 (3.3)
Time until treatment [Mean (Standard Deviation); unit: hour] | 7.7 (5.9) | 7.6 (3.6) | 5.6 (3.0) | 7.0 (4.2)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 148.6 (14.6) | 150.7 (13.7) | 152.5 (12.8) | 150.6 (13.7)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 88.7 (10.7) | 85.1 (13.6) | 87.2 (12.5) | 87.0 (12.3)
National Institutes of Health Stroke Scale score [Mean (Standard Deviation); unit: units on a scale] — The scores range from 0 to 42, with higher scores indicating increasing severity. A score of < 4 represented low-degree impairment, between 4 and 15 represented medium-degree impairment, and a score of > 15 represented severe-degree impairment.
  units on a scale | 12.4 (4.38) | 10.6 (4.74) | 10.2 (3.72) | 11.1 (4.28)
Barthel Index score [Mean (Standard Deviation); unit: units on a scale] — The scores range from 0, indicating complete dependence on help with activities of daily living, to 100, indicating independence.
  units on a scale | 19.75 (6.38) | 22.25 (7.16) | 22.00 (6.96) | 21.33 (6.83)

OUTCOME MEASURES:

1. Primary Outcome: National Institutes of Health Stroke Scale Score
Description: Scores range from 0 to 42, with higher scores indicating increasing severity
Time Frame: At 11-day and 21-day after therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dl-3-n-butylphthalide | Cerebrolysin | Placebo
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Day 11 | 8.78 (2.48) | 7.80 (5.81) | 8.85 (4.43)
  Day 21 | 5.48 (2.34) | 5.90 (3.96) | 7.30 (4.78)

2. Secondary Outcome: Barthel Index Score
Description: Range from 0, indicating complete dependence on help with activities of daily living, to 100, indicating independence
Time Frame: At 11-day and 21-day after therapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dl-3-n-butylphthalide | Cerebrolysin | Placebo
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  Day 11 | 35.25 (10.57) | 36.00 (10.81) | 31.00 (8.68)
  Day 21 | 54.00 (14.01) | 53.75 (13.10) | 43.75 (15.50)

ADVERSE EVENTS:
Time Frame: 21 days
Description: Systematic methods include a physical examination (including heart rate, blood pressure and oxygen concentration), laboratory tests (including urine test, complete blood count, occult blood test, renal function, liver function, electrolyte and blood-glucose), electrocardiogram, cranial CT or MRI and chest radiograph.
Arm/Group | Dl-3-n-butylphthalide | Cerebrolysin | Placebo
Serious Adverse Events (participants affected / at risk) | 8/20 | 7/20 | 11/20
Other Adverse Events (participants affected / at risk) | 16/20 | 12/20 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dl-3-n-butylphthalide (N=20) | Cerebrolysin (N=20) | Placebo (N=20)
Coagulation disorder (Blood and lymphatic system disorders) | 6 (10) | 3 (6) | 5 (8)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 4 (5)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dl-3-n-butylphthalide (N=20) | Cerebrolysin (N=20) | Placebo (N=20)
Erythrema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Fever (General disorders) | 5 (9) | 3 (5) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 3 (5)
Nausea/vomiting (General disorders) | 4 (7) | 2 (5) | 2 (6)
Anemia (Blood and lymphatic system disorders) | 5 (7) | 4 (6) | 2 (4)

LIMITATIONS AND CAVEATS:
Foremost is the relatively small sample size, and only patients with moderate severity of stroke were enrolled, so the efficacy results of this study should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes